CLINICAL TRIAL: NCT05541276
Title: MELAtonin for Prevention of Postoperative Agitation and Emergence Delirium in Children. The MELA-PAED Trial: a Randomized, Double-blind, Placebo-controlled Trial.
Brief Title: MELAtonin for Prevention of Postoperative Agitation and Emergence Delirium in Children
Acronym: MELA-PAED
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Sygehus Lillebaelt (Other); University of Copenhagen (Other); Copenhagen Trial Unit, Center for Clinical Intervention Research (Other)
Responsible Party: Principal Investigator, Arash Afshari, Head of Research, Associated Professor, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 20211125; 2021-006464-24 (EudraCT Number)
Record Dates: First submitted 2022-09-12; First posted 2022-09-15 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Emergence Delirium
Keywords: Anesthesia; Melatonin; Sevoflurane; Postoperative Pain; Child; PONV
MeSH Terms: conditions — Emergence Delirium; Pain, Postoperative; Postoperative Nausea and Vomiting | interventions — Melatonin; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Melatonin (Experimental): Participants receive melatonin solution for injection 1 mg/mL in a dosage of 0.15 mg/kg body weight as a single intravenous injection approximately 30 minutes before end of surgical procedure.
  Interventions: Drug: Melatonin
- Placebo (Placebo Comparator): Participants receive isotonic sodium chloride (9mg/mL) intravenously once approximately 30 minutes before end of surgical procedure in a volume equivalent to the melatonin group for the same weight.
  Interventions: Drug: Isotonic sodium chloride solution

INTERVENTIONS:
Drug: Melatonin — Melatonin for injection 1 mg/mL
  Arms: Melatonin
Drug: Isotonic sodium chloride solution — Sodium chloride 0.9 % for injection
  Other Names: Normal saline
  Arms: Placebo

SUMMARY:
Postoperative agitation and emergence delirium describe a spectrum of symptoms of early postoperative negative behavior, in which the child experiences a variety of behavioral disturbances including crying, thrashing, and disorientation during early awakening from anaesthesia. The symptoms are common with a reported incidence of approximately 25%. Some clinical trials have studied the effect of prophylactic oral melatonin for reducing the risk of emergence agitation in children, some finding a considerable dose-response effect. Melatonin has a low bio-availability of approximately 15 %. The safety of exogenous melatonin for pediatric patients has been studied with no apparent serious adverse effects, even at repeated short-term use of high doses of intravenous melatonin. The aim of this clinical trial is to investigate the prophylactic effects and safety of intravenous melatonin administered intraoperatively for prevention of postopreative agitation and emergence delirium in children after an elective surgical procedure. The study is designed as a randomised, double-blind, placebo-controlled clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 1-6 years
* Elective surgical procedure of en axpected duration of at least 30 minutes in general anesthesia maintained with sevoflurane

Exclusion Criteria:

* Any known allergy or contraindication to study treatment or excipåients
* Current daily medication with melatonin

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 400 (Estimated)
Dates: Start 2025-01-21 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of emergence agitation | Up to approximately 4 hours corresponding to stay in Post-Anesthetic Care Unit (PACU).
  Participants will be assessed on Watcha scale repeatedly ever 15 min during their stay at the Post-Anesthetic Care Unit. The variable is dichotomous: any score >2= "Yes" and no score <=2 = "No"

SECONDARY OUTCOMES:
Opioid consumption | Up to approximately 4 hours corresponding to stay in Post-Anesthetic Care Unit (PACU).
  The total amount of opioids administered for postoperative pain in the PACU will be evaluated as units of morphine equivalents per kg. No more than 35 % of the popu-lation is expected to receive postoperative opioids in a range of approximately 10-100 µg/kg.
Non-serious Adverse Events (AE) | From enrolment to the trial until 24-hour follow-up.
  Any untoward medical occurrence not considered serious.

OTHER OUTCOMES:
Serious Adverse Events (SAE) | SAEs will be assessed from enrolment until 30 days after intervention.
  We will use the International Conference on Harmonization of technical require-ments for registration of pharmaceuticals for human use-Good Clinical Practice (ICH-GCP) definition of a serious adverse event, which is any untoward medical occurrence that resulted in death, was life-threatening, re-quired hospitalization or prolonging of existing hospitalization and resulted in persistent or significant disability or jeopardized the participant.
Postoperative pain | Up to approximately 4 hours corresponding to stay in Post-Anesthetic Care Unit (PACU).
  The incidence of postoperative pain will be assessed in each group according to the FLACC scale, assessed every 15 minutes in PACU. Postoperative pain is defined as any FLACC score >3.
Postoperative nausea and vomiting (PONV) | Up to approximately 4 hours corresponding to stay in Post-Anesthetic Care Unit (PACU).
  The incidence of PONV will be assessed dichotomously every 15 minutes in PACU. Outcome assessors will observe for vomiting. Nausea can be considered present if the participant refuses to eat and other causes are ruled out. There is no adequate PONV assessment tool available. PONV will be considered present if any assess-ment during PACU stay is "Yes".
Time to administration of opioid | Up to approximately 4 hours corresponding to stay in Post-Anesthetic Care Unit (PACU).
  Time from end of anesthesia to the time point at which the first dose of opioid is administered in PACU. Not all participants (expectedly up to approximately 35%) will receive opioids in PACU.
Need for rescue medication | Up to approximately 4 hours corresponding to stay in Post-Anesthetic Care Unit (PACU).
  Dichotomous assessment of any administration in PACU of rescue medication specifically targeting EA according to treatment algorithm i.e., clonidine or propofol.
Time to awakening in PACU | Up to approximately 4 hours corresponding to stay in Post-Anesthetic Care Unit (PACU).
  Time from end of anesthesia to the first time point at which the participant is awake. If the participant is not awake two hours after arrival in PACU, a wake-up at-tempt will be carried out.
Time to postoperative oral intake | Up to approximately 4 hours corresponding to stay in Post-Anesthetic Care Unit (PACU).
  Time from end of anesthesia to the first time point at which the participant eats/drinks. All participants are assumed to eat/drink during their PACU stay.
Time for discharge readiness | Up to approximately 4 hours corresponding to stay in Post-Anesthetic Care Unit (PACU).
  Time from end of anesthesia (defined as above) to the time point at which partici-pant fulfills local discharge criteria. Discharge criteria will be evaluated by the re-sponsible physician prior to final discharge from PACU either to the participant's ward or to their home.
Emergence delirium | Up to approximately 4 hours corresponding to stay in Post-Anesthetic Care Unit (PACU).
  The incidence of emergence delirium will be evaluated according to the PAED score assessed every 15 minutes during PACU stay. The end-point is defined dichotomously as any score ≥10. Due to feasibility concerns, this outcome will solely be evaluated in a sub-population of approximately 50% of the trial population (200 participants), specifically only thos enrolled at the Juliane Marie Center Site.
Readmissions within 30 days | From day of discharge + 30 days.
  Assessed dichotomously counting day 0 as the day of discharge from hospital after the procedure. For the small group (expectedly <5 %) who will have had any read-missions within 30 days, the number of readmissions will be described.

CONTACTS AND LOCATIONS:
Overall Officials: Arash L Afshari, MD, PhD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Department of Anesthesiology, Juliane Marie Center, Rigshospitalet, Copenhagen, Capital Region, Denmark